CLINICAL TRIAL: NCT06312189
Title: Open-Label Study of Valbenazine for the Treatment of Chorea Associated With Huntington Disease in Canada
Brief Title: Long-term Study to Evaluate Safety and Tolerability of Valbenazine in Participants With Chorea Associated With Huntington Disease in Canada
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Neurocrine Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NBI-98854-HD3022
Record Dates: First submitted 2024-03-08; First posted 2024-03-15 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Chorea, Huntington
MeSH Terms: conditions — Huntington Disease | interventions — valbenazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Valbenazine (Experimental): Capsule, administered orally once daily.
  Interventions: Drug: Valbenazine

INTERVENTIONS:
Drug: Valbenazine — vesicular monoamine transporter 2 (VMAT2) inhibitor
  Other Names: NBI-98854

SUMMARY:
This study will evaluate long-term safety and tolerability of valbenazine in participants with chorea associated with Huntington Disease (HD) who participated in Study NBI-98854-HD3006 (NCT04400331) in Canada.

ELIGIBILITY:
Key Inclusion Criteria:

* Participated in Study NBI-98854-HD3006 and completing dosing through the Week 156 visit; or were actively participating, receiving study treatment, and completed an early termination visit Study NBI-98854-HD3006 at the time of the study closure at sites in Canada.
* Participants of childbearing potential must agree to use contraception consistently while participating in the study until 30 days after last dose of the study treatment.

Key Exclusion Criteria:

* Have difficulty swallowing
* Are currently pregnant or breastfeeding
* Have a medically significant abnormality, physical examination finding, clinically significant laboratory abnormality

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Estimated)
Dates: Start 2024-04-24 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment-Emergent Adverse Events (TEAEs) | Up to Week 106

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Lead, Study Director — Neurocrine Biosciences
Locations (3):
- Canada (3):
  - Neurocrine Clinical Site, Vancouver, British Columbia
  - Neurocrine Clinical Site, Ottawa, Ontario
  - Neurocrine Clinical Site, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No